CLINICAL TRIAL: NCT05209672
Title: The Relationship Between the Global Limb Anatomic Staging System (GLASS) and Short Term Outcomes of Endovascular Management of Infrainguinal Lesions in Patients With Chronic Limb Threatening Ischemia (CLTI)"
Brief Title: GLASS Classification and CLTI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ahmed Shawki Roshdi, Responsible investigator, Assiut University
Other Study IDs: GLASS
Record Dates: First submitted 2021-12-13; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Chronic Limb-Threatening Ischemia Nos of Native Arteries of Extremities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Critical limb threatening ischemia "CLTI 'is not a separate local disease but also it is a part of generalized vascular disorder. A clinical syndrome that can be presented by many symptoms and signs as rest pain, gangrene and chronic ulceration more than 2 weeks (1).

DETAILED DESCRIPTION:
The Global Vascular guidelines 'GVG "proposes a new Global Anatomic Staging System (GLASS), GLASS incorporates two novel and important concepts, the target arterial path (TAP) and estimated limb-based patency (LBP). Based on appropriate angiographic imaging, the TAP is defined by the treating surgeon or internationalist as the optimal arterial pathway to restore in-line (pulsatile) flow to the ankle and foot. LBP allows more direct comparison of anatomic outcomes across revascularization strategies in CLTI. The complexity of disease traversed by the TAP is integrated in the GLASS. Femoropopliteal (FP) and infrapopliteal (IP) arterial segments are individually graded on a scale of 0 to 4.(2)(3) Using a consensus based matrix, these segmental grades are combined into three overall GLASS (I-III) stages for the limb, reflecting the complexity of the disease with a proposed likelihood of immediate technical failure ' ITF " and 1 year "LBP " after endovascular intervention of " TAP ' (1)

ELIGIBILITY:
Inclusion Criteria:

* Patients with infrainguinal CLTI

Exclusion Criteria:

* Patients with concomitant Aorto-iliac lesions
* Acute ischemia patients
* Post Traumatic ischemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending the Vascular Surgery Clinics in Assiut University Hospitals with infra inguinal CLTI will be recruited to participate in the study. Based on high quality angiography, patients presented with CLTI will be assigned into 3 stages according to GLASS
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Imitate technical failure | 1 year
  Failure of passage of wire or Recoil of vessels during angioplasty
Limb based patency at 1 year | 1 year
  Patent vessels after endovascular management

SECONDARY OUTCOMES:
Amputation free survival at 1 year | 1 year
  Limb preserved after endovascular intervention
Mortality Rate at 1 year | 1 year
  Death after endovascular intervention
Amputation rate at 1 year | 1 year
  Amputation after endovascular intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Conte MS, Bradbury AW, Kolh P, White JV, Dick F, Fitridge R, Mills JL, Ricco JB, Suresh KR, Murad MH, Aboyans V, Aksoy M, Alexandrescu VA, Armstrong D, Azuma N, Belch J, Bergoeing M, Bjorck M, Chakfe N, Cheng S, Dawson J, Debus ES, Dueck A, Duval S, Eckstein HH, Ferraresi R, Gambhir R, Gargiulo M, Geraghty P, Goode S, Gray B, Guo W, Gupta PC, Hinchliffe R, Jetty P, Komori K, Lavery L, Liang W, Lookstein R, Menard M, Misra S, Miyata T, Moneta G, Munoa Prado JA, Munoz A, Paolini JE, Patel M, Pomposelli F, Powell R, Robless P, Rogers L, Schanzer A, Schneider P, Taylor S, De Ceniga MV, Veller M, Vermassen F, Wang J, Wang S; GVG Writing Group for the Joint Guidelines of the Society for Vascular Surgery (SVS), European Society for Vascular Surgery (ESVS), and World Federation of Vascular Societies (WFVS). Global Vascular Guidelines on the Management of Chronic Limb-Threatening Ischemia. Eur J Vasc Endovasc Surg. 2019 Jul;58(1S):S1-S109.e33. doi: 10.1016/j.ejvs.2019.05.006. Epub 2019 Jun 8. PMID 31182334